CLINICAL TRIAL: NCT05755490
Title: PROWESS (PROstate Cancer Wearables Exercise and Structured Supports): A Pilot Supportive Care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel E Lage, MD, MSc, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-609
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: Prostate Cancer; Prostatic Neoplasms; Androgen Deprivation Therapy; ADT; CBR; Cognitive Behavioral Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Yohimbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PROWESS (Experimental): Participants will complete study procedures as outlined:
  * Wear FitBit watch during the 12-week study period.
  * Group intervention sessions, in-person or virtually.
  * One optional follow-up session.
  * One-on-one, semi-structured interview with trained study staff to assess participant experience with intervention.
  Interventions: Behavioral: PROWESS

INTERVENTIONS:
Behavioral: PROWESS — Structured, culturally sensitive behavior change intervention comprised of six video-based or in-person sessions with psychologist or social worker. FitBit is provided by study.

SUMMARY:
The goal of this research study is to conduct an open pilot of a behavioral change intervention called PROstate Cancer Wearables, Exercise, and Structured Supports (PROWESS) for integrating health behavior change tools and to increase exercise, reduce side effects of androgen deprivation therapy (ADT), and improve quality of life in Black and Hispanic/Latino men with prostate cancer.

The name of the intervention used in this research study is:

PROWESS (behavioral change intervention)

DETAILED DESCRIPTION:
This research study is to test a behavioral change intervention called PROstate Cancer Wearables, Exercise, and Structured Supports (PROWESS) for integrating health behavior change tools with wearable technology, to increase exercise, reduce side effects of androgen deprivation therapy (ADT), and improve quality of life in Black and Hispanic/Latino men with prostate cancer on androgen deprivation therapy (ADT).

Study procedures include screening for eligibility, intervention sessions, questionnaires and surveys, and an exit interview with study staff.

Participation in this research study is expected to last for up to four months.

The goal and primary outcome of this open pilot study is refinement of the intervention and study procedures to allow for us to conduct a larger feasibility study in the future.

It is expected that about 10 people will take part in this research study.

This research study is being supported by the MGH Cancer Center

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer.
* Planning to be on androgen deprivation therapy (ADT) for at least three months
* Black Race AND/OR Hispanic/Latino Ethnicity (confirmed by patient self-report)
* Verbal fluency in English or Spanish.
* Receiving ongoing oncology care at MGH Cancer Center.
* Age ≥ 18 years.
* Self-Report less than or equal to 150 minutes of moderate or vigorous structured exercise per week, as assessed by the Exercise is Medicine Physical Activity Vital Sign Assessment
* Completion of baseline assessment

Exclusion Criteria:

* Unwilling or unable to participate in the study.
* Significant psychiatric, cognitive or other comorbid disease which the treating clinician believes prohibits informed consent or participation in the study.
* Currently receiving chemotherapy.
* Prognosis less than 6 months, per the judgment of the primary oncologist.
* Medical contraindication to physical activity, as assessed by outpatient oncologist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Participant Satisfaction | At week 8-12 (intervention completion)
  Assessed by the Client Satisfaction Questionnaire-3 (CSQ), a 3-item survey with answers ranging from 1-4, "quite dissatisfied" to "very satisfied."

SECONDARY OUTCOMES:
Change in Objective Physical Activity | At Baseline and from weeks 1 - 12
  Collected physical activity via FitBit measure of steps and activity classification.
Change in Self-Reported Exercise | At Baseline and weeks 8-12
  Assessed by the Short-Form International Physical Activity Questionnaire (IPAQ), a self-reported measure of physical activity.
Change in Participant Quality of Life | At Baseline and weeks 8-12
  Assessed by the Functional Assessment of Cancer Therapy-Prostate (FACT-P), which consists of five subscales assessing physical, functional, emotional, social wellbeing.
Change in Psychological Distress Symptoms | At Baseline and weeks 8-12
  Assessed by the Patient Health Questinnaire-4, a 4-item measure with two separate subscales to evaluate symptoms of anxiety and depression.
Change in Self-Efficacy for Managing Symptoms | At Baseline and weeks 8-12
  Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions - Managing Symptoms Scale, an 8-item measure to evaluate self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lage, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation